CLINICAL TRIAL: NCT00393406
Title: The Influence of Breast Cancer Risk and Risk Perception on Lifestyle Behaviors Among Women With a Family History: A Mixed Method Approach
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907013; 07-E-N013
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-28

CONDITIONS: Breast Neoplasms
Keywords: Objective Risk; Gail Model; Subjective Risk; Medical Risk-Reducing Strategies; Physical Activity, Diet, Alcohol Use; Breast Cancer Risk
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Alcohol Drinking

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Lifestyle behaviors among women with a family history of breast cancer are likely to be influenced by a number of factors, including both objective risk factors and subjective risk, or perceived risk. The aims of this mixed method study are twofold and will be explored through both quantitative (i.e. secondary survey data) and qualitative data (i.e. personal in-depth interviews) derived from the Sister Study, a large epidemiologic study being conducted through the National Institute of Environmental Health Sciences, which is addressing risk factors for breast cancer in sisters of women who have had breast cancer. The quantitative aims include an exploration of lifestyle behaviors and behavioral differences between White and African American women, as well as well as an exploration of the relationships between lifestyle behaviors (i.e. varying levels of objective risk based on Gail model risk scores, medical risk-reducing factors (i.e. use of Tamoxifen or Raloxifene and/or prophylactic surgery), as well as additional factors that may be contributors to perceived risk. This aim will be addressed using data that have already been collected as part of the baseline activities for the Sister Study. The primary qualitative aim is to gain a better understanding about perceived risk and the relationship between perceived risk and lifestyle behaviors in both White and African American women with a family history of breast cancer. This aim requires the collection of new data through in-person interviews with between 28 and 40 women, depending on how many interviews are required to achieve "data saturation."

The mixed method approach will be based on a "complementarity" model, which emphasizes the use of two different methods to address different aspects of the research problem. Results from both methods will become integrated into the discussion of the findings and it is expected that this approach will enrich the study and allow for elaboration of the quantitative results. The secondary data analysis will be derived from approximately 10,000 women, initially enrolled in the Sister Study, who are between the ages of 35 and 74 and have had at least one sister affected by breast cancer. Women for the qualitative interviews will be recruited from a cohort of Sister Study participants residing within North Carolina and will include equal numbers of both White and African American women. It is expected that 28 women will be needed for qualitative data saturati...

DETAILED DESCRIPTION:
Lifestyle behaviors among women with a family history of breast cancer are likely to be influenced by a number of factors, including both objective risk factors and subjective risk, or perceived risk. The aims of this mixed method study are twofold and will be explored through both quantitative (i.e. secondary survey data) and qualitative data (i.e. personal in-depth interviews) derived from the Sister Study, a large epidemiologic study being conducted through the National Institute of Environmental Health Sciences, which is addressing risk factors for breast cancer in sisters of women who have had breast cancer. The quantitative aims include an exploration of lifestyle behaviors and behavioral differences between White and African American women, as well as an exploration of the relationships between lifestyle behaviors (i.e. varying levels of objective risk based on Gail model risk scores, medical risk-reducing factors (i.e. use of Tamoxifen or Raloxifene and/or prophylactic surgery), as well as additional factors that may be contributors to perceived risk. This aim will be addressed using data that have already been collected as part of the baseline activities for the Sister Study. The primary qualitative aim is to gain a better understanding about perceived risk and the relationship between perceived risk and lifestyle behaviors in both White and African American women with a family history of breast cancer. This aim requires the collection of new data through in-person interviews with between 28 and 40 women, depending on how many interviews are required to achieve "data saturation."

The mixed method approach will be based on a "complementarity" model, which emphasizes the use of two different methods to address different aspects of the research problem. Results from both methods will become integrated into the discussion of the findings and it is expected that this approach will enrich the study and allow for elaboration of the quantitative results. The secondary data analysis will be derived from approximately 10,000 women, initially enrolled in the Sister Study, who are between the ages of 35 and 74 and have had at least one sister affected by breast cancer. Women for the qualitative interviews will be recruited from a cohort of Sister Study participants residing within North Carolina and will include equal numbers of both White and African American women. It is expected that 28 women will be needed for qualitative data saturation (i.e. no new information comes forth) to occur.

The primary outcome measures for the quantitative component of the study are dietary fat intake, fruit and vegetable consumption, alcohol use and physical activity, which will all be measured categorically. Physical activities will first be converted into MET (metabolic equivalent) values and then MET values will be summed across all activities before categorizing into quartiles or quintiles. Qualitative data will be analyzed through content analysis, which will involve the identification of common themes or ideas expressed in response to questions from a semi-structured interview guide developed specifically to address the aims of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Data from the first 20,000 women enrolled in the Sister Study will be utilized for the quantitative analysis.

Participants for the qualitative study will include women living in North Carolina who reside within a three and a half hour driving distance from the researcher.

EXCLUSION CRITERIA:

The only exclusion criteria for the selection of data from women in the Sister Study are as follows:

1. women will be excluded if they were adopted because a complete family history is unlikely to be known;
2. women will be excluded if they have had prior history of cancer, with the exception of non-melanoma skin cancer;
3. women from racial/ethnic groups classified as "other" will also be excluded.

The same exclusion criteria described above will also apply for the qualitative study.

Ages: 35 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-10-24; Study Completion 2008-10-28

CONTACTS AND LOCATIONS:
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Aiken LS, Fenaughty AM, West SG, Johnson JJ, Luckett TL. Perceived determinants of risk for breast cancer and the relations among objective risk, perceived risk, and screening behavior over time. Womens Health. 1995 Spring;1(1):27-50. PMID 9373372
- [Background] Ainsworth BE, Haskell WL, Leon AS, Jacobs DR Jr, Montoye HJ, Sallis JF, Paffenbarger RS Jr. Compendium of physical activities: classification of energy costs of human physical activities. Med Sci Sports Exerc. 1993 Jan;25(1):71-80. doi: 10.1249/00005768-199301000-00011. PMID 8292105
- [Background] Audrain J, Lerman C, Rimer B, Cella D, Steffens R, Gomez-Caminero A. Awareness of heightened breast cancer risk among first-degree relatives of recently diagnosed breast cancer patients. The High Risk Breast Cancer Consortium. Cancer Epidemiol Biomarkers Prev. 1995 Jul-Aug;4(5):561-5. PMID 7549815